CLINICAL TRIAL: NCT06214429
Title: Evaluation of Atherosclerotic Carotid Plaque Stiffness by Shear Wave Elastography, Greyscale Median, Magnetic Resonance Imaging and Histopathological Analysis: Diagnostic Test Study
Brief Title: Shear Wave Elastography for Carotid Atherosclerotic Plaques
Status: Recruiting | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Principal Investigator, Matheus Bertanha, PhD, Professor, UPECLIN HC FM Botucatu Unesp
Other Study IDs: UPECLIN-MB-7
Record Dates: First submitted 2023-12-28; First posted 2024-01-19 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Carotid Atherosclerosis
MeSH Terms: conditions — Carotid Artery Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carotid Atherosclerotic Plaque Stenosis >50%: Main cohort, composed by subjects with carotid stenosis above 50% confirmed by at least methods (eg. Doppler ultrasound peak systolic velocity > 140cm/s and MRI residual lumen measurement).
  Interventions: Diagnostic Test: Vascular Ultrasound; Diagnostic Test: Shear Wave Elastography; Diagnostic Test: Greyscale Median; Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: Histopathology

INTERVENTIONS:
Diagnostic Test: Vascular Ultrasound — Complete vascular ultrasound routine in B mode, color mode and Doppler.
Diagnostic Test: Shear Wave Elastography — Vascular ultrasound assisted shear wave elastography of the atherosclerotic plaque.
Diagnostic Test: Greyscale Median — Vascular ultrasound assisted assessment of the plaque in B mode. The plaque image will be post-processed for the histogram median value for the plaque area.
Diagnostic Test: Magnetic Resonance Imaging — Assessment of the plaque and carotid residual lumen by magnetic resonance.
Diagnostic Test: Histopathology — Histopathology findings for patients that undergo carotid endarterectomy.

SUMMARY:
The goal of this prospective diagnostic accuracy cohort study is to compare the accuracy of carotid atherosclerotic plaques stiffness assessed by shear wave elastography (SWE) with greyscale median values (GSM), magnetic resonance imaging (MRI) and histopathological findings in patients with carotid atherosclerotic plaques causing stenosis above 50%, symptomatic or not.

The main question it aims to answer is: is the plaque stiffness correlatable with GSM values, MRI findings or histopathological findings? Participants will be subjected to a vascular ultrasound study in which the SWE and GSM will be assessed. The second imaging modality for stenosis confirmation will be MRI and patients with confirmed symptomatic stenosis above 50% or assymptomatic stenosis above 70% will be considered for surgery intervention (endarterectomy or angioplasty). Patients that undergo endarterectomy will have the carotid plaques subjected to a histopathological study. The study will not arbitrate about the treatment decision.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atherosclerotic carotid plaques that develop stenosis superior to 50%.

Exclusion Criteria:

* Previous cervical surgery;
* Previous cervical radiotherapy;
* Stenosis caused by vascular inflammatory diseases;
* Pregnant women;
* High carotid bifurcation (inaccessible by vascular ultrasound linear probe);
* Posterior acoustic shadowing that impair morphological evaluation of the plaque.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of outpatient care subjects referred to the Noninvasive Vascular Laboratory of the Hospital das Clinicas da Faculdade de Medicina de Botucatu for vascular appointments or vascular ultrasound assessment for carotid atherosclerotic disease.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Plaque Stiffness | Through study completion, an average of 2 years.
  Measured in kilopascal (kPa).
Plaque Greyscale | Through study completion, an average of 2 years.
  Median value of plaque histogram.
Plaque Instability (MRI) | Through study completion, an average of 2 years.
  Degree of plaque instability as proposed by American Heart Association (I to IV).
Plaque Instability (Histopathology) | If patient is submitted to carotid endarterectomy.
  Degree of plaque instability as proposed by American Heart Association (I to IV).

SECONDARY OUTCOMES:
Plaque Surface | Through study completion, an average of 2 years.
  Regular, irregular or calcified.
Anatomic Site of Stenosis | Through study completion, an average of 2 years.
  Common carotid artery, bifurcation, internal carotid artery, external carotid artery.
Plaque Correlation with Arterial Wall | Through study completion, an average of 2 years.
  Concentric or eccentric.
Fibrotic Cap | Through study completion, an average of 2 years.
  Thin, thick or absent.
Echolucent Plaque Area | Through study completion, an average of 2 years.
  Present or absent.
Plaque Echogenicity | Through study completion, an average of 2 years.
  Echolucent, predominantly echolucent, predominantly echogenic, echogenic or calcified.
Ulceration | Through study completion, an average of 2 years.
  Present or absent.
Peak Systolic Velocity | Through study completion, an average of 2 years.
  At the site of highest velocity and turbulent flow in centimeters per second (cm/s).
End Diastolic Velocity | Through study completion, an average of 2 years.
  At the site of highest velocity and turbulent flow in centimeters per second (cm/s).
Velocity Ratio | Through study completion, an average of 2 years.
  At the site of highest velocity and turbulent flow compared to ipsilateral pre-stenosis common carotid artery.
ECST Morphological Degree of Stenosis | Through study completion, an average of 2 years.
  Percentage of stenosis as measured by the European Carotid Surgery Trial (ECST) protocol (%).
NASCET Morphological Degree of Stenosis | Through study completion, an average of 2 years.
  Percentage of stenosis as measured by the The North American Symptomatic Carotid Endarterectomy Trial (NASCET) protocol (%).

CONTACTS AND LOCATIONS:
Overall Officials: Matheus Bertanha, Ph.D., Study Chair — São Paulo State University
Locations (1):
- Sao Paulo State University, Botucatu, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No